CLINICAL TRIAL: NCT06449105
Title: The Effect of Mindfulness Compassionate Life Practice on Stress, Self-Efficacy and Quality of Life in Hemodialysis Patients: A Randomized Controlled Study
Brief Title: The Effect of Mindfulness Compassionate Living Practice on Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mine CENGİZ, Lecturer doctor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCENGİZ3
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Hemodialysis Patients
Keywords: Hemodialysis patients; Mindfulness; Life quality; Self-Efficacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Session 1: How We Evolved - Threat, Impulse, and Soothing Systems (Experimental): •A "breath break with kindness" is practiced. •Encourage them to think about how threat, impulse and sedative systems have developed in their own lives. •A "safe place" application is made. • "Courtesy meditation" is done.
  Interventions: Behavioral: 1: How We Evolved - Threat, Impulse, and Soothing Systems
- Session 2: Threat and Self-Compassion (Experimental): •A "breath break with kindness" is practiced. • "Building a compassionate relationship with resilience" and "kindness meditation: a benevolent" practices are made. • "A hand on your heart" and "a compassionate comrade" practices are made.
  Interventions: Behavioral: Session 2: Threat and Self-Compassion
- Session 3: Unraveling the Knots of Desire and Patterns Agenda (Experimental): •Talk about homework. •A "breath break with kindness" is practiced. • "Establishing a compassionate relationship with desire", "guided meditation to discover the inner pattern", "courtesy meditation: a good friend" practices are made.
  Interventions: Behavioral: Session 3: Unraveling the Knots of Desire and Patterns Agenda
- Session 4: Internalizing compassion (Experimental): • "Pretend-to-pretend" practice is made for participants to observe themselves. • In addition to the previous practices, the practice of "internalizing compassion" is made in order to increase their expanded mindfulness. •Courtesy meditation: a neutral person", "kindness towards your body", which is based on mindfulness practices and increases body awareness and mindful movement, is carried out. During the day, they will be informed that they should do the "walking with kindness" practice on their own
  Interventions: Behavioral: Session 4: Internalizing compassion
- Session 5: Me and others - Expanding the circle (Experimental): •A "compassionate letter" application is made by asking participants to think about a situation they encountered recently or some time ago and is still causing distress. It is explained that they can gain insight with this application. • "Courtesy meditation: the 'difficult' person", "compassion and breathing: yourself" and "compassionate breathing: others" practices are made
  Interventions: Behavioral: Session 5: Me and others - Expanding the circle
- Session 6: Growing happiness (Experimental): • "Revisiting the good" practice is carried out to define the five sense organs for the participants. • "Forgiveness", "Asking for forgiveness", "forgiving others", "gratitude" practices are carried out. •The practice is expanded as "kindness meditation: groups and all beings".
  Interventions: Behavioral: Session 6: Growing happiness
- : Session 7: Weaving Wisdom and Compassion into Daily Life (Experimental): •Participants are made to choose a day in their life and allow a few minutes to pause in a mindful way. • "A breather for wise and compassionate action", "calmness meditation" and "joy sharing meditation" practices are carried out.
  Interventions: Behavioral: Session 7: Weaving Wisdom and Compassion into Daily Life
- Session 8: Living with the Heart (Experimental): •The participants are told about the applications that they can apply for, where they need help to develop compassion towards self-healing skills, and the whole training is evaluated. •The "river of life" application, which evaluates mindfulness in depth, is carried out. •An overall summary of the 8-session study is made and feedback is received.
  Interventions: Behavioral: Session 8: Living with the Heart

INTERVENTIONS:
Behavioral: 1: How We Evolved - Threat, Impulse, and Soothing Systems — The practice of "Breath break with kindness" will be applied for 5 minutes. Afterwards, 15 minutes of information on threats, impulses and soothing systems, "A safe place" application for 11 minutes, "Courtesy meditation" for 10 minutes. After each application, 10 minutes of feedback will be received from the participants.
  Arms: Session 1: How We Evolved - Threat, Impulse, and Soothing Systems
Behavioral: Session 2: Threat and Self-Compassion — The practice of "breathing with kindness" will be done for 7 minutes. The practice of "Building a compassionate relationship with resilience" will be held for 12 minutes, and the practice of "Kindness meditation: a benevolent" will take place for 11 minutes. "A hand over your heart" application will be made for 3 minutes and "A compassionate comrade" application will be done for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 2: Threat and Self-Compassion
Behavioral: Session 3: Unraveling the Knots of Desire and Patterns Agenda — The practice of "breathing with kindness" will be done for 7 minutes. "Building a compassionate relationship with desire" 12 minutes, "Guided meditation to discover the inner pattern" 10 minutes and "Courtesy meditation: a good friend" 11 minutes. Except for the "breath break with kindness" application, 3 minutes of feedback will be received from the participants after each application
  Arms: Session 3: Unraveling the Knots of Desire and Patterns Agenda
Behavioral: Session 4: Internalizing compassion — The "pretend-to-be" practice for the participants to observe themselves will be made for 10 minutes. The practice of "internalizing compassion" will be done for 7 minutes, "kindness meditation: a neutral person" practice for 10 minutes, and "kindness towards your body" for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 4: Internalizing compassion
Behavioral: Session 5: Me and others - Expanding the circle — The "a compassionate letter" practice with the participants will continue for 15 minutes. "meditation: the 'difficult' person" 8 minutes, "compassion and breathing: yourself" 10 minutes and "compassionate breathing: others" 7 minutes. A "compassionate break" application is performed for 7 minutes.
  Arms: Session 5: Me and others - Expanding the circle
Behavioral: Session 6: Growing happiness — The practice of "Revisiting the good" is carried out for 10 minutes with the participants. "Forgive yourself", "wish for forgiveness", "forgive others", "gratitude" practices will be held for 5 minutes each and will take 20 minutes in total. "Courtesy meditation: groups and all beings" will be practiced for 10 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: Session 6: Growing happiness
Behavioral: Session 7: Weaving Wisdom and Compassion into Daily Life — Participants will be given 10 minutes to choose a day in their life and allow a few minutes to pause mindfully. The practice of "a breather for wise and compassionate action" is 10 minutes, the practice of "calmness meditation" is 8 minutes, and the practice of "sharing the joy meditation" is 8 minutes. After each application, 3 minutes of feedback will be received from the participants.
  Arms: : Session 7: Weaving Wisdom and Compassion into Daily Life
Behavioral: Session 8: Living with the Heart — The participants are told about the applications they can apply for, where they need help to develop compassion towards self-healing skills, and the entire training will be evaluated for 20 minutes. The "river of life" application is carried out for 20 minutes. 10 minutes of feedback will be received after the application.
  Arms: Session 8: Living with the Heart

SUMMARY:
There are studies evaluating the effects of mindfulness-based practices on individuals receiving HD treatment. No studies have been found on how Mindfulness Compassionate Life application reduces stress, increases self-efficacy and quality of life in individuals receiving HD treatment. Considering the stress situations experienced by individuals receiving HD treatment, it is thought that the evidence-based effect of Mindfulness Compassionate Living application on individuals' stress, self-efficacy and quality of life is important.

The population of the research will consist of 90 Hemodialysis patients who were treated in Bingöl State Hospital Dialysis Unit during the specified date range. Sample size of the research; Calculated using the GPower computer program. With the power analysis, it was calculated that at the α = 0.05 level, the effect size would be strong 150, 153 (d = 0.8) and the power of the study would be 90%, and that at least 68 patients should be included in the sample. Patients who meet the research criteria and agree to participate in the research will be randomly assigned to one experimental and one control group.

DETAILED DESCRIPTION:
Introductory information form prepared by the researcher in line with the literature and containing the socio-demographic data of hemodialysis patients, Perceived Stress Scale (PSS) to evaluate stress, Self-Efficacy-Efficacy Scale (SEES) to evaluate self-efficacy, SF-12 Quality of Life Scale to evaluate quality of life. , Self-Compassion Scale Short Form (PSS-K) will be used to evaluate self-compassion, and Conscious Mindfulness Scale (BIPS) will be used to evaluate conscious mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with chronic renal failure
* Being over 18 years of age,
* Being willing to participate in the study
* Being open to communication and collaboration

Exclusion Criteria:

* Having a diagnosis of acute renal failure,
* Having a current hospital stay,
* Lack of openness to communication and collaboration,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | up to 1 day
  The form consists of 14 questions containing information about the patient treated in the dialysis unit, created by the researcher within the scope of the literature. The created form includes questions regarding the patient's age, gender, educational status, marital status, number of children (if any), economic status and disease process.

SECONDARY OUTCOMES:
Perceived Stress Scale | up to 1 day
  It was developed by Cohen, Kamarck and Mermelste in 1983 to determine the perceived stress level of participants. The scale was adapted to Turkish by Bilge, Öğce, Genç and Oran (2007), and the Cronbach alpha value was found to be 0.82 in the reliability study. In the scale, some situations that include the feelings and thoughts that individuals may have experienced during the past month are given. Individuals marked the situation in each item by thinking about how much they lived during the last month. The scale is five-point Likert type. A high total score means a high level of perceived stress. In the reliability study of the scale, Cronbach's alpha value was found to be 0.86.

OTHER OUTCOMES:
Self-Efficacy Scale | up to 1 day
  Developed by Sherer and Madduks in 1982, ÖEYÖ was adapted into Turkish by Gözüm and Aksayan in 1999. ÖEYÖ is a 5-point Likert type self-assessment scale. The scale has 23 items and four subgroups, for each item; It is required to mark one of the options: 1."Does not describe me at all", 2."Describes me a little", 3."I am undecided", 4."Describes me well", 5."Describes me very well". A minimum of 23 and a maximum of 115 points can be obtained from the scale. A high total score from the scale indicates that the individual's perception of SEE is at a good level.
Quality of Life Index-Dialysis III Version | up to 1 day
  The Turkish validity and reliability study of the scale, which was developed by Ferrans and Powers in 1987, was conducted by Korkut in 2007. The Cronbach alpha reliability coefficient of the scale is 0.90 (20). The scale consists of two different sections expressing satisfaction and importance and each section consists of 34 items. With a total of 68 items and six-point Likert-type items, in the satisfaction section, from "very satisfied" to "very dissatisfied"; and in the importance part, the answers are given from "very important" to "very unimportant". Additionally, there are four sub-dimensions in each section: health and function, socio-economic, psychological-beliefs and family dimension.
Self-Compassion Scale Short Form | up to 1 day
  The Turkish validity and reliability of the scale developed by Neff (2003) was conducted by Yıldırım and Sarı in 2018. It has been confirmed that the scale has a structure consisting of 11 items, a single dimension, and two complementary components (positive component and negative component). The internal consistency coefficient of the scale was calculated as .75. PSQ-K is recommended to be used in studies that will use total scores to measure self-compassion.
Mindful Awareness Scale | up to 1 day
  It was developed by Brown and Ryan27 for the purpose of evaluating individuals' BF level. In the validity and reliability study of the scale conducted on a university sample in Turkey, the Cronbach alpha coefficient was found to be 0.80.28 The scale is a one-dimensional, six-point Likert type evaluation scale consisting of 15 questions. The minimum and maximum score that individuals can get from the scale is between 15 and 90. High scores indicate high BF level.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Cengiz, Principal Investigator — Atatürk University, Faculty of Nursing